CLINICAL TRIAL: NCT02408705
Title: A Randomized, Double Blind, Two-period Cross-over Trial Investigating the Effect of Liraglutide as Add on to Intensive Insulin Treatment on the Endogenous Glucose Production in Subjects With C-peptide Positive Type 1 Diabetes Mellitus
Brief Title: Investigating the Effect of Liraglutide on the Endogenous Glucose Production During in Tye 1 Diabetes Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of Graz (Other)
Collaborators: Novo Nordisk A/S (Industry)
Responsible Party: Principal Investigator, Pieber Thomas, MD, Univ.Prof. Dr., Medical University of Graz
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: LG_T1_EGP
Record Dates: First submitted 2015-01-28; First posted 2015-04-03 (Estimated); Last update posted 2016-09-12 (Estimated); Status verified 2016-09

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Endogenous Glucose Production; Hypoglycemic clamp; Tracer to Tracee Technique; Type 1 diabetes mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Liraglutide; Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Liraglutide (Active Comparator): 3-month treatment of liraglutide
  Interventions: Drug: Liraglutide; Drug: Mixed Meal Tolerance Test with paracetamol
- Placebo (Placebo Comparator): 3-month treatment of placebo
  Interventions: Drug: Placebo; Drug: Mixed Meal Tolerance Test with paracetamol

INTERVENTIONS:
Drug: Liraglutide — They are receiving liraglutide for 3 months. Dose escalation: 0.3 mg - 0.6mg - 0.9mg - 1.2mg (over 4 weeks)
  Other Names: Victoza
  Arms: Liraglutide
Drug: Placebo — They are receiving placebo for 3 months. Dose escalation: 0.3 mg - 0.6mg - 0.9mg - 1.2mg (over 4 weeks)
  Arms: Placebo
Drug: Mixed Meal Tolerance Test with paracetamol — At the beginning and end of each period (Visit 2a, 8, 9a, 15) a Mixed Meal Tolerance Test enriched paracetamol will be performed.
  Other Names: MMTT

SUMMARY:
Each subject will be allocated to 2 periods of 3 months of once daily dosing with either liraglutide (1.2 mg) or placebo treatment (in random sequence) as add on to usual intensive insulin treatment. Wash-out period between treatments will be 1 month.

The trial can be divided into the following periods:

* Screening
* Treatment period 1
* Washout period
* Treatment period 2
* Follow up Visit

Mixed Meal Tolerance Test (MMTT) enriched with paracetamol:

At the beginning and end of each period a MMTT (Fortimel complete) enriched with paracetamol will be performed to assess the remaining beta-cell function via obtained maximal plasma C-peptide levels as well as the gastric emptying.

Experimental / Hypoglycaemic clamp :

At the end of each period (Visit 8, 15) a hypoglycaemic clamp will be performed. After the subject completed the MMTT on day 1, the subject will stay in the clinical unit to prepare for the hypoglycaemic clamp with an variable insulin infusion intravenously in order to obtain a steady state of a plasma glucose (PG) level of 5.5 mmol/L overnight until approximately 08:00. At 05:00 hours 10%-[6,6-2H2] glucose solution will be given i.v. as a primed (9.6mg/kg/min) for one minute and a constant (0.08 mg/kg/min) infusion until the last blood sampling of the plateau 4.0 mmol/L will be performed.

At 08:00 hours in the morning at day 2, insulin infusion will be increased to 1.5 mU/kg/min for each subject and the PG will be kept at a plateau of 5.5 mmol/L by a controlled variable intravenous infusion of glucose (10% glucose enriched with 4mg [6,6-2H2] glucose /ml) for one hour. Afterwards, PG is allowed to fall to a plateau of 3.5 mmol/L, then to a nadir of 2.5 mmol/L, then to a blood glucose of 4.0 mmol/L and finally back to a level of 5.5 mmol/L for safety reasons. Blood sampling for measurement of [6,6-2H2] glucose, glucagon, insulin, counterregulatory hormones, lactate, free fatty acids, glycerol, vital signs, hypoglycaemic symptoms questionnaire and hypoglycaemic awareness will be performed at each PG plateau.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent obtained before any trial-related activities. Trial-related activities are any procedures that are carried out as part of the trial, including activities to determine suitability for the trial
2. Type 1 diabetes mellitus as diagnosed (including I - III):

   I. history of type 1 diabetes mellitus manifestation with acute hyperglycaemia and ketonuria II. positive results for at least one of four islet antibodies (glutamic acid decarboxylase, protein tyrosine phosphatase, zinc transporter 8, or islet cell antibodies) III. residual basal fasting C-peptide of ≥ 0.1 nmol/L
3. Male or female, aged 18 - 64 years (both inclusive)
4. Body mass index (BMI) 20.0 - 25.0 kg/m2 (both inclusive)
5. HbA1c 42 - 80 mmol/mol (6.0-9.5%)
6. Treated with daily insulin injections or continuous s.c. insulin infusion (CSII) ≥ 1 months. Stable insulin dose as judged by the investigator

Exclusion Criteria:

1. Known or suspected hypersensitivity to trial product(s) or related products
2. Use of liraglutide or exenatide within 3 months before screening
3. Severe hypoglycaemia within 1 month of screening
4. Hypoglycaemia unawareness as judged by the Investigator or hospitalisation for diabetic ketoacidosis during the previous 2 months
5. Clinically significant abnormal haematology, biochemistry, lipids, or urinalysis or coagulation screening tests, as judged by the investigator and any of the following laboratory safety results:

   * Aspartate transaminase(=AST), alanine aminotransferase (=ALT), lipase, alkaline phosphatase > 2.0 times upper limit of reference range (ULN)
   * Haemoglobin < 8.0 mmol/L (male) or < 6.4 mmol/L (female), total leukocyte count <3.0 x 109/L, thrombocytes <100 x 109/L
   * Serum creatinine levels ≥ 126 μmol/L (male) or ≥ 111 μmol/L (female)
   * Amylase outside normal range
6. Screening calcitonin > 50 ng/L
7. Personal history of non-familial medullary thyroid carcinoma
8. History of chronic or idiopathic acute pancreatitis Suffer from or history of a life threatening disease (e.g. cancer except basal cell skin cancer or squamous cell skin cancer), or any clinically significant respiratory, metabolic, renal, hepatic, gastrointestinal, endocrinological (with the exception of diabetes mellitus and euthyroid struma), haematological, dermatological, venereal, neurological, psychiatric diseases or other major disorders as judged by the investigator.
9. Proliferative retinopathy or maculopathy and/or severe neuropathy, in particular autonomic neuropathy, as judged by the investigator.
10. Any disease or condition that, in the opinion of the investigator, would represent an unacceptable risk for the subject's safety.
11. Any condition that would interfere with trial participation or evaluation of results, as judged by the investigator.
12. Female of child-bearing potential who is pregnant, breast-feeding or intend to become pregnant or is not using adequate contraceptive methods (adequate contraceptive methods include sterilisation, hormonal intrauterine devices, oral contraceptives, sexual abstinence or vasectomised partner).
13. Severe acute and/or chronic diseases

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2015-01; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Area under the curve of the endogenous glucose production from (=EGP) from begin of the hypoglycaemic clamp 5.5 mmol/L period until the end of recovery period (4.0 mmol/L), calculated from stable isotope labelled plasma glucose | After 12 weeks and 2 days of treatment in each treatment period (day 86 and day 198)

SECONDARY OUTCOMES:
Area under the curve of peripheral glucose uptake (=PGU), calculated from labelled PG from begin of the hypoglycaemic clamp period 5.5mmol/L until end of recovery period (4.0 mmol/L) | After 12 weeks and 2 days of treatment in each treatment period (day 86 and day 198)
Area under the glucose infusion rate curve from begin of the hypoglycaemic clamp period 5.5mmol/L until end of recovery period (4.0 mmol/L) | After 12 weeks and 2 days of treatment in each treatment period (day 86 and day 198)
Change in mean plasma glucagon concentrations from begin of the hypoglycaemic clamp period 5.5 mmol/L to 3.5 mmol/L to nadir and to recovery phase | After 12 weeks and 2 days of treatment in each treatment period (day 86 and day 198)
Change in mean values of adrenaline from begin of the hypoglycaemic clamp period 5.5 mmol/L to 3.5 mmol/L to nadir and to recovery phase | After 12 weeks and 2 days of treatment in each treatment period (day 86 and day 198)
Change in mean values of noradrenaline from begin the hypoglycaemic clamp period 5.5 mmol/L to 3.5 mmol/L to nadir and to recovery phase | After 12 weeks and 2 days of treatment in each treatment period (day 86 and day 198)
Change in mean values of cortisol from begin the hypoglycaemic clamp period 5.5 mmol/L to 3.5 mmol/L to nadir and to recovery phase | After 12 weeks and 2 days of treatment in each treatment period (day 86 and day 198)
Change in mean values of growth hormone from begin the hypoglycaemic clamp period 5.5 mmol/L to 3.5 mmol/L to nadir and to recovery phase | After 12 weeks and 2 days of treatment in each treatment period (day 86 and day 198)
Change in number of regulatory T-cells detected by blood (fasting) and measured by a laboratory | After 12 weeks and 2 days of treatment just before the hypoglycaemic clamp in each treatment period (day 86 and day 198)
Change in function of regulatory T-cells detected by blood (fasting) and measured by a laboratory | After 12 weeks and 2 days of treatment just before the hypoglycaemic clamp in each treatment period (day 86 and day 198)
Area under the glucose curve during the Mixed Meal Tolerance Test | Period 1: Visit 2a (Day 1) versus Visit 8 (Day 85) ; Period 2: Visit 9a (Day 113) versus Visit 15 (Day 197)
Area under the c-peptid concentration curve during the Mixed Meal Tolerance Test | Period 1: Visit 2a (Day 1) versus Visit 8 (Day 85) ; Period 2: Visit 9a (Day 113) versus Visit 15 (Day 197)
Area under the paracetamol concentration curve to calculate gastric emptying during the Mixed Meal Tolerance Test | Period 1: Visit 2a (Day 1) versus Visit 8 (Day 85) ; Period 2: Visit 9a (Day 113) versus Visit 15 (Day 197)
Area under the insulin curve during the Mixed Meal Tolerance Test | Period 1: Visit 2a (Day 1) versus Visit 8 (Day 85) ; Period 2: Visit 9a (Day 113) versus Visit 15 (Day 197)
Area under the glucagon curve during the Mixed Meal Tolerance Test | Period 1: Visit 2a (Day 1) versus Visit 8 (Day 85) ; Period 2: Visit 9a (Day 113) versus Visit 15 (Day 197)
Change in HbA1c during each period detected by blood (fasting) at the begin of the visits and measured by a laboratory (tube: K3 EDTA Plasma) | Period 1: Visit 2a (Day 1) versus at Visit 8 (Day 85) ; Period 2: Visit 9a (Day 113) versus Visit 15 (Day 197)
Change in fasting plasma glucose during each period detected by blood at the begin of the visits and measured by a laboratory (tube: lithium heparin plasma) | Period 1: Visit 2a (Day 1) versus Visit 8 (Day 85) ; Period 2: Visit 9a (Day 113) versus Visit 15 (Day 197)

OTHER OUTCOMES:
Number of treatment emergent adverse events | From begin of the trial (Day 1) until the end of the trial (Day 204)
Number of self-reported hypoglycaemic episodes during each period | Day 1 until Day 86 (Period 1) compared with Day 113 until day 198 (Period 2)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas R. Pieber, MD, Principal Investigator — Medical University of Graz
Locations (1):
- Medical University Graz, Graz, Austria

REFERENCES:
- [Derived] Zenz S, Regittnig W, Boulgaropoulos B, Augustin T, Brunner M, Korsatko S, Munzker J, Narath SH, Raml R, Magnes C, Pieber TR. Effect of Liraglutide Treatment on Whole-body Glucose Fluxes in C-peptide-Positive Type 1 Diabetes During Hypoglycemia. J Clin Endocrinol Metab. 2022 Aug 18;107(9):e3583-e3593. doi: 10.1210/clinem/dgac369. PMID 35833597
- See also: Medical University of Graz — http://www.medunigraz.at